CLINICAL TRIAL: NCT07276607
Title: The Effect of Nada Yoga Music and Stress Ball Use on Anxiety and Pain Levels During Smear Smear Tests in Women: A Randomized Controlled Trial
Brief Title: The Effect of Nada Yoga Music and Stress Ball Use on Anxiety and Pain Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, nurten özçalkap, Asistant Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/73
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Intervention Effectiveness
Keywords: Pain; anxiety; nada yoga music; pap smear; stress ball
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This research was a prospective, parallel, randomized controlled trial with pretest, posttest, and follow-up measurements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Nada Yoga Music
  Interventions: Other: Nada Yoga Music
- Group 2 (Experimental): Stress Ball
  Interventions: Other: Stress Ball group:
- Group 3 (Experimental): Nada Yoga Music + Stress Ball
  Interventions: Other: Nada Yoga Music + Stress Ball group
- Group 4 (No Intervention): standard care group

INTERVENTIONS:
Other: Nada Yoga Music — Participants listened to Nada Yoga music through headphones for 15 minutes before and 15 minutes after the Pap smear procedure.
  Arms: Group 1
Other: Stress Ball group: — Participants were instructed to perform squeeze-release exercises using a medium-firm stress ball during the procedure.
  Arms: Group 2
Other: Nada Yoga Music + Stress Ball group — Participants both listened to Nada Yoga music and performed stress ball exercises concurrently.
  Arms: Group 3

SUMMARY:
This parallel-group randomized controlled trial was conducted between Aprıl 2025 and December 2025 at a Training and Research Hospital in Türkiye among women who applied for Pap smear testing. A total of 128 participants aged 30-56 years were included. Data were collected at three time points using the Personal Information Form, Visual Analog Scale (VAS), and State-Trait Anxiety Inventory (STAI). A mixed-model ANOVA was applied to address the effects of time, group, and time × group interactions. Statistical significance was set at p≤0.05.

DETAILED DESCRIPTION:
The study population consisted of women who applied for a Pap smear test at X Training and Research Hospital between Aprıl 2025 and December 2025 . The sample size was calculated using the G*Power 3.1.9.7 software (Faul et al., 2007). Based on a medium effect size (0.25), a two-way mixed-design ANOVA (repeated measures, within-between interaction), an alpha error of 0.05, an inter-measurement correlation of 0.5, and a statistical power of 95% (1-β = 0.95), the minimum required sample size was determined to be 60 (15 per group). The study was completed with a total of 128 voluntary participants, distributed equally across four groups: Nada Yoga Music (n = 32), Stress Ball (n = 32), Nada Yoga Music + Stress Ball (n = 32), and Control (n = 32). The inclusion criteria included being between 30 and 65 years of age, having no communication barriers, applying for a Pap smear test, and volunteering to participate in the study. The exclusion criteria included having any condition preventing music listening (e.g., hearing loss), having any limitation preventing stress ball use (e.g., hand or finger injuries), or having a diagnosed psychiatric disorder (e.g., depression, bipolar disorder).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included being between 30 and 65 years of age, having no communication barriers, applying for a Pap smear test, and volunteering to participate in the study

Exclusion Criteria:

* The exclusion criteria included having any condition preventing music listening (e.g., hearing loss), having any limitation preventing stress ball use (e.g., hand or finger injuries), or having a diagnosed psychiatric disorder (e.g., depression, bipolar disorder).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Average 8 Years
  It is a form prepared by the researcher based on the relevant literature to assess the sociodemographic characteristics of the participants.
Visual Analog Scale | Average 8 Years
  The Visual Analogue Scale (VAS) was first developed in 1921 by Hayes and Patterson. The standard VAS, as generally accepted, is a semi-quantitative, ordinal scale consisting of a 100-mm line. This scientifically accepted standard length aims to provide an easy and quantitative method of assessment. The VAS was first used as a self-rated tool to measure mood in 1969 by Zealley and Aitken.
  Studies conducted with VAS in patients experiencing pain have shown that the horizontal format is used more frequently. The VAS is typically defined as a 10-cm line, either horizontal or vertical, starting with "No Pain" and ending with "Unbearable Pain." This line may be presented as a simple straight line or divided into equal segments. When used to assess pain, it may also include descriptive pain labels placed along the line.
  The VAS has been a successful assessment tool in many studies for determining the effects of treatment. In our study, participants were asked to indicate their pain level o
Spielberger State Anxiety Inventory | Average 8 Years
  Spielberger's State-Trait Anxiety Inventory (STAI):
  Developed in 1964 by Spielberger et al., the State-Trait Anxiety Inventory was designed to measure the state and trait anxiety levels of both normal and clinical populations. The scale was adapted into Turkish by Öner and Le Compte. It is a self-report instrument composed of brief statements. The State Anxiety Inventory (SAI) provides information only about how the individual feels at that specific moment, whereas the Trait Anxiety Inventory (TAI) was developed to assess anxiety experienced over the past seven days.
  The STAI consists of two subscales, each containing 20 items, rated on a 4-point Likert scale. In a study conducted with both healthy and clinical samples, Aydemir and Köroğlu (2000) reported reliability coefficients ranging from .83 to .87.

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Özçalkap, Principal Investigator — AĞRI İBRAHİM ÇEÇEN UNIVERSTY; SİBEL YÜCETÜRK, Study Chair — SİNOP UNIVERSTY
Locations (1):
- Ağri İbrahim Çeçen Universty, Ağrı, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283